CLINICAL TRIAL: NCT05809791
Title: Prevalence and Clinical Characteristics of Molar Incisor Hypomineralization (MIH) and Hypomineralized Second Primary Molars (HSPM) Among Italian, Spanish and Turkish Children: a Multicenter Epidemiological Study
Brief Title: Molar Incisor Hypomineralization and Hypomineralized Second Primary Molars
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 11/21
Record Dates: First submitted 2023-03-28; First posted 2023-04-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization (MIH); Hypomineralized Second Primary Molars (HSPM); Prevalence
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Molar and Incisor Hypomineralization (MIH) is a qualitative developmental defect of the dental enamel with a multifactorial aetiology defined in 2001 as an "hypomineralization of systemic origin affecting one or more permanent molars, usually first permanent molars (FPMs) with or without the involvement of one or more affected permanent incisors". Due to its porous structure with an altered prism organization and an increased content of proteins, the hypomineralized enamel has reduced mechanical properties and a lower refractive index in comparison to the sound enamel. MIH is associated to a large number of objective and subjective problems as an altered aesthetics, an increased risk of plaque accumulation, caries and/or post-eruptive breakdown, reduced retention rates of adhesive materials, hypersensitivity and difficulty in anesthetizing the affected teeth that make its management a challenging condition. MIH is a very widespread pathology with a worldwide prevalence ranging from 2.8 to 44% and a global average prevalence of 13.1% with significant geographical differences. In 2015, the number of global prevalent cases was estimated at 878 million people with a percentage of needing-care cases of 27.4% (in mean 240 million prevalent cases). In Europe, MIH prevalence rates between 3.6 to 25%. Regarding Italy, a limited number of prevalence studies are available. Recently, literature reports that the presence of MIH-like lesions in primary dentition, especially on second primary molars, may be a predictive factor for developing MIH in permanent dentition. However, the absence of this defect called Hypomineralized Second Primary Molars (HSPM) does not rule out MIH development. The early diagnosis of HSPM is very useful to early diagnose MIH and reduce its care burden. The reported HSPM global prevalence rate ranges from 0 to 21.8% with a global average about 7.88%. MIH and HSPM are both very widespread pathologies affecting an increasing number of children worldwide and represent a significant problem in pediatric dentistry. The aim of this study is to estimate the prevalence of MIH in Italian (Trieste), Spanish (Huesca, Zaragoza) and Turkish (Istanbul) children. The hypothesis is that the estimated prevalence of MIH may be in line with that reported in literature and that the presence of HSPM in primary dentition may be associated with MIH development in permanent dentition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-16 years;
* Signature of the informed consent to the study by patients' parents or by their legal guardians

Exclusion Criteria:

* Fluorosis, white spots, amelogenesis imperfecta, hypoplasia or other dental enamel defects in differential diagnosis with MIH and HSPM;
* Patients not sufficiently cooperative;
* Children with orthodontic devices hiding the teeth to consider

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be selected among patients attending the involved Dental Clinics according to the following criteria
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
MIH prevalence rate | At baseline (day one)
  Prevalence of the condition in the populations studied

SECONDARY OUTCOMES:
Description of MIH clinical characteristics | At baseline (day one)
  Description of the clinical characteristics of MIH, evaluated by questionnaire
Frequency of the most frequently affected teeth | At baseline (day one)
  Evaluated by questionnaire
Association between HSPM and MIH development | At baseline (day one)
  Evaluated by questionnaire
Association between MIH/HSPM and presence of caries | At baseline (day one)
  Evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Milena Cadenaro, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (5):
- Italy (3):
  - IRCCS Burlo Garofolo, Trieste, Italy
  - Maggiore Hospital, Trieste, Trieste
  - IRCCS Burlo Garofolo, Trieste
- Servicio de Odontología de la Universidad de Zaragoza, Huesca, Huesca, Spain
- Faculty of Dentistry of the Yeditepe University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No